CLINICAL TRIAL: NCT06779747
Title: Evaluation of Different Diagnostic Therapeutic Strategies in Patients with Thyroid Pathology
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: TirBo
Record Dates: First submitted 2024-12-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-11

CONDITIONS: Hypothyroidism; Hyperthyroidism/Thyrotoxicosis; Thyroid Nodule (Benign); Thyroid Carcinoma
MeSH Terms: conditions — Hypothyroidism; Hyperthyroidism; Thyrotoxicosis; Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective Group: The retrospective phase will involve about 2850 patients of whom:
  * 500 with hypothyroidism;
  * 500 suffering from hyperthyroidism/thyrotoxicosis;
  * 1000 affe8ed with benign thyroid nodule;
  * 850 suffering from thyroid carcinoma.
- Prospective Group: In the prospective phase, on the other hand, about 3000 patients will be sequentially enrolled, including:
  * 60/year with hypothyroidism;
  * 60/year suffering from hyperthyroidism/thyrotoxicosis;
  * 100/year suffering from benign thyroid nodule;
  * 80/year suffering from thyroid carcinoma.

SUMMARY:
Observational single-center prospective and retrospective, nonpharmacological, spontaneous cohort study.

DETAILED DESCRIPTION:
The study is observational single-center prospective and retrospective, nonpharmacological, spontaneous cohort study. This study will be offered to any patient with thyroid pathology (hypothyroidism, hyperthyroidism/thyrotoxicosis, benign thyroid nodule, and thyroid carcinoma) followed by our Center with a minimum 3-month follow-up. In the retrospective phase, patients in whom thyroid pathology was diagnosed from 01/01/1995 until the approval of this study will be enrolled, while in the prospective phase those diagnosed from the time of the approval of this study to the next 10 years will be enrolled. In both phases, each patient will be followed for a maximum duate of 20 years.

Patients participating in the study will not undergo any procedure (laboratory or instrumental examination, examination or treatment) that is beyond the scope of normal daily clinical practice. Likewise, the clinical variables that will be collected for the study are those that are commonly collected by the physician in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years at the time of diagnosis;
* Patients with thyroid pathology (hypothyroidism, hyperthyroidism/thyrotoxicosis, benign thyroid nodule, and thyroid carcinoma) in whom the diagnosis was made in our Center or another Center from 01/01/1995 until the approval of this study (retrospective phase) or from the time of approval of this study to the next 10 years (prospective phase);
* Obtaining informed consent.

Exclusion Criteria:

* Follow up lasting less than 3 months;
* Incomplete or missing clinical data that may affect the correct assessment of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with thyroid pathology (hypothyroidism, hyperthyroidism/thyrotoxicosis, benign thyroid nodule, and thyroid carcinoma) followed at our Center with a minimum 3-month follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 5850 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2041-12-29 (Estimated); Study Completion 2041-12-30 (Estimated)

PRIMARY OUTCOMES:
Characterization of Patient Population with Thyroid Disease (Hypothyroidism, Hyperthyroidism, Benign Nodules, Thyroid Carcinoma) | through study completion, an average of 17 years
  The primary objective is to describe the characteristics of the patient population followed at our Center for any thyroid disease (hypothyroidism, hyperthyroidism/thyrotoxicosis, benign thyroid nodule, and thyroid carcinoma), through specific data collection, with the intent to improve their clinical-diagnostic-therapeutic management.

SECONDARY OUTCOMES:
Comparison of L-Thyroxine Formulations (Capsules, Soft-Gel, Liquid) in Hypothyroidism Therapy | through study completion, an average of 17 years
  This measure will compare the clinical and laboratory improvements in hypothyroidism therapy with different formulations of L-thyroxine (capsules, soft-gel, liquid). The improvements will be assessed based on changes in thyroid function tests (e.g., TSH, T4 levels) and related clinical symptoms.
Comparison of L-Thyroxine + L-Thyronine Combination Therapy in Hypothyroidism | through study completion, an average of 17 years
  This measure will evaluate the clinical-laboratory improvements in hypothyroidism therapy using a combination of L-thyroxine and L-thyronine. The assessment will focus on changes in thyroid function (e.g., TSH, T4) and patient-reported outcomes, such as fatigue and quality of life.
Evaluation of Drug-Induced Dysthyroidism | through study completion, an average of 17 years
  This measure will assess drug-induced dysthyroidisms (hypothyroidism and hyperthyroidism) caused by various drugs, including thyrotosteroids, iodine excess, lithium, amiodarone, INF, immunomodulators, and TKIs. The assessment will include clinical evaluations and thyroid function tests (e.g., TSH, T4) to monitor drug-related thyroid changes.
Impact of the Great Score on Radio-Metabolic Therapy Response in Basedow's Disease | through study completion, an average of 17 years
  This outcome measure will evaluate the prognostic impact of the Great Score and other factors in predicting the response to radio-metabolic therapy in patients with Basedow's disease. The primary assessment will include clinical response measures such as thyroid function tests and symptom resolution.
Evaluation of Efficacy and Adverse Effects of Local or Systemic Drugs in Basedow's Ophthalmopathy and Pretibial Myxedema | through study completion, an average of 17 years
  This measure will assess the efficacy and adverse effects of local or systemic drug treatments in Basedow's ophthalmopathy and pretibial myxedema. Evaluations will include changes in symptoms (e.g., ocular signs, skin changes) and any treatment-related adverse effects.
Evaluation of Prognostic Impact of the McGill Score for Cytologically Indeterminate Thyroid Nodules | through study completion, an average of 17 years
  This outcome measure will evaluate the prognostic impact of the McGill Score in patients with cytologically indeterminate thyroid nodules. The outcome will focus on predicting malignancy risk using the McGill Score, as well as other factors, and will include follow-up biopsy and surgical outcomes.
Evaluation of Additional Prognostic Factors for Malignancy in Thyroid Nodules | through study completion, an average of 17 years
  This measure will evaluate additional prognostic factors for malignancy in thyroid nodules, including molecular markers, imaging characteristics, and other clinical factors. These will be assessed in combination with the McGill Score to predict malignancy risk.
Efficacy and Adverse Effects of Minimally Invasive Treatments for Thyroid Nodules (Radiofrequency, Laser) | through study completion, an average of 17 years
  This outcome measure will evaluate the efficacy and adverse effects of minimally invasive treatments (e.g., radiofrequency ablation, laser therapy) for thyroid nodules. The assessment will include changes in nodule size, symptoms, and any procedure-related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Uberto Pagotto, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No